CLINICAL TRIAL: NCT01282827
Title: Paraorbital-occipital Alternating Electric Current Stimulation in Patients With Optic Neuropathy
Brief Title: Paraorbital-Occipital Electric Stimulation in Patients With Optic Neuropathy (BCT_optnerve)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Magdeburg (Other)
Collaborators: EBS Technologies GmbH (Industry)
Responsible Party: Principal Investigator, Bernhard A. Sabel, Director, Inst Med Psychol, University of Magdeburg
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EBS-optnerv-BCT
Record Dates: First submitted 2011-01-21; First posted 2011-01-25 (Estimated); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Visual Impairment
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- rtACS (Verum condition) (Experimental): Repetitive transorbital alternating current stimulation (rtACS)
  Interventions: Device: rtACS (verum condition)
- Placebo stimulation (Placebo Comparator): no intervention (Sham stimulation)
  Interventions: Device: placebo stimulation

INTERVENTIONS:
Device: rtACS (verum condition) — Repetitive, transorbital alternating current stimulation (rtACS) was applied with a multi-channel device generating weak current pulses in predetermined firing bursts of 2 to 9 pulses. The amplitude of each current pulse was below 1000 microA. Current intensity was individually adjusted according to how well patients perceived phosphenes, i.e. any sensation of flickering light in response to the rtACS stimulation.
  Other Names: Device for electrical stimulation "Brainstim"; Hersteller: "ELSTIM", St. Petersburg, Russland; Device number: "07062006"; Classification: Class II, Type BF; SLG device marking: "5016-07-P/001"; Modifications of the device have been performed before the SLG test by "Eurotronics Weißenfelser Straße 67, D-04229 Leipzig"
  Arms: rtACS (Verum condition)
Device: placebo stimulation — a clicking sound was presented and the same electrodes montage set-up was used during rtACS and placebo stimulation, except that placebo patients received no current (stimulator turned off).
  Other Names: Device for electrical stimulation "Brainstim"; Hersteller: "ELSTIM", St. Petersburg, Russland; Device number: "07062006"; Classification: Class II, Type BF; SLG device marking: "5016-07-P/001"; Modifications of the device have been performed before the SLG test by "Eurotronics Weißenfelser Straße 67, D-04229 Leipzig"
  Arms: Placebo stimulation

SUMMARY:
Non-invasive brain stimulation can increase cortical excitability in the visual system, but it is not known if this is of clinical value. The investigators now assessed if repetitive, transcranial alternating current stimulation (rtACS) can improve visual field size in patients with optic nerve damage. The investigators hypothesized that rtACS would improve visual functions with the defective visual field sectors of the visual field (primary outcome measure).

DETAILED DESCRIPTION:
exploratory, randomized, controlled study

ELIGIBILITY:
Inclusion Criteria:

* residual vision
* patients with optic nerv lesion
* lesion age at least 6 months
* stable visual field defect

Exclusion Criteria:

* electric or electronic implants such as pace maker
* any metal artefacts in head and truncus
* epilepsia
* photosensitive epilepsy as determines by EEG
* autoimmune illnesses in acute stage
* mental diseases such e.g. schizophrenia etc.
* diabetes causing diabetic retinopathy
* addiction
* high blood pressure
* unstable or high level intraocular pressure (i.e. > 27 mmHg)
* retinitis pigmentosa
* pathological nystagmus
* presence of an un-operated tumor or tumor recidive

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Detection accuracy (DA) change in percent over baseline within defective visual field sectors | between baseline and 60 days after stimulation
  Central visus fields were assessed with computer based high-resolution perimetry (HRP). Based on such plots, areas of the visual field were characterized as intact, partially damaged or absolutely impaired (blind).

SECONDARY OUTCOMES:
Visual Parameters 1 | baseline to 60 days after stimulation
  DA in static and kinetic perimetry
Visual Parameters 2 | baseline to 60 days after stimulation
  reaction time (RT) in HRP
Visual Parameters 3 | baseline to 60 days after stimulation
  visual acuity (VA)
Visual Parameters 4 | baseline to 60 days after stimulation
  contrast vision
EEG parameters | baseline to 60 days after stimulation
  EEG power spectra

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard A Sabel, Prof. Dr., Principal Investigator — University of Magdeburg
Locations (2):
- Germany (2):
  - Klinik für Neurologie, Charité Campus Mitte, Universitätsmedizin Berlin, Berlin
  - Institut für Medizinische Psychologie, Leipziger Str. 44, Magdeburg